CLINICAL TRIAL: NCT06612346
Title: Minimally Invasive Nasal Trabeculostomy: Long-Term Follow-Up Extension Study
Status: Completed | Type: Observational
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MMS-EEU-7
Record Dates: First submitted 2024-08-27; First posted 2024-09-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Open Angle Glaucoma
Keywords: MINT; Trabeculostomy; Minimally Invasive Glaucoma Surgery; MIGS; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINT Surgery Cohort: Cohort that includes subjects that have undergone the MINT surgical procedure.
  Interventions: Device: Minimally Invasive Micro Trabeculostomy

INTERVENTIONS:
Device: Minimally Invasive Micro Trabeculostomy — The MINT system is a surgical device designed to create a trabeculostomy within the eye.
  Other Names: MINT

SUMMARY:
This study is a follow-up extension study conducted in continuation of the prior MINT study (MMS-EEU-4), in which the long-term (i.e., 18, 24 months) clinical outcomes of Minimally Invasive Nasal Trabeculostomy (MINT) will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years to ≤ 85 years old
2. Subject who underwent MINT, and surgery was performed not earlier than 18 months from enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects of Armenian descent that underwent the MINT procedure.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure Measurement | 18 months +/- 2 months post-MINT surgery from previous study (MMS-EEU-4).
  Observed IOP at long-term timepoints

OTHER OUTCOMES:
Adverse Events Outcomes | 0-24 +/-2 months post MINT surgery from previous study (MMS-EEU-4).
  Incidence of adverse events related to MINT device/procedure, including visual acuity and postoperative complications, throughout the study follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- S. Malayan Eye Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided